CLINICAL TRIAL: NCT05971810
Title: Perioperative Oral Decontamination and ImmunoNuTrition (POINT) on Postoperative Pulmonary Complications in Elderly: a Multicenter Randomized Controlled Trial
Brief Title: Perioperative Oral Decontamination and ImmunoNuTrition (POINT) in Elderly
Acronym: POINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Fujian Provincial Hospital (Other); The Second Hospital of Hebei Medical University (Other); Shenzhen Qianhai Shekou Free Trade Zone Hospital (Unknown); Ningbo No.2 Hospital (Other); Peking University International Hospital (Other); Guizhou Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: I-23PJ953
Record Dates: First submitted 2023-07-21; First posted 2023-08-02 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Complications; Pulmonary Complication
Keywords: immunonutrition; oral decontamination; postoperative pulmonary complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (immunonutrition and oral chlorhexidine decontamination, IN&CD) (Experimental): Patients in this group will receive immunonutrition supplementation from the day of allocation at the preoperative anesthesia clinic until the day before surgery (usually 1-3 weeks), which is oral intake of ORAL IMPACT™ 2 servings per day. Patients will also receive oral chlorhexidine decontamination using 0.12% chlorhexidine oral rinse twice daily from the day before surgery until postoperative day 3.
  Interventions: Dietary Supplement: immunonutrition supplement of ORAL IMPACT™; Other: oral chlorhexidine decontamination
- Group B (immunonutrition and routine oral care, IN&RC) (Experimental): Patients in this group will receive immunonutrition supplementation from the day of allocation at the preoperative anesthesia clinic until the day before surgery (usually 1-3 weeks), which is oral intake of ORAL IMPACT™ 2 servings per day. For oral health care, they will receive routine oral care which is routine toothbrushing twice daily.
  Interventions: Dietary Supplement: immunonutrition supplement of ORAL IMPACT™
- Group C (routine nutrition advice and oral chlorhexidine decontamination, RN&CD) (Experimental): Patients in this group will be advised to follow a standard nutrition advice with a total intake of 30kcal/kg/d and protein intake of 1.2g/kg/d. They will also receive oral chlorhexidine decontamination using 0.12% chlorhexidine oral rinse twice daily from the day before surgery until postoperative day 3.
  Interventions: Other: oral chlorhexidine decontamination
- Group D (routine nutrition advice and routine oral care, RN&RC) (No Intervention): Patients in this group will be advised to follow a standard nutrition advice with a total intake of 30kcal/kg/d and protein intake of 1.2g/kg/d. They will also receive routine oral care which is routine toothbrushing twice daily.

INTERVENTIONS:
Dietary Supplement: immunonutrition supplement of ORAL IMPACT™ — For intervention group, patients will take immunonutrition supplement after recruitment until the day before surgery.
  Arms: Group A (immunonutrition and oral chlorhexidine decontamination, IN&CD); Group B (immunonutrition and routine oral care, IN&RC)
Other: oral chlorhexidine decontamination — For intervention group, patients will use 0.12% chlorhexidine for oral rinse twice daily from the day before surgery until 3 days after surgery.
  Arms: Group A (immunonutrition and oral chlorhexidine decontamination, IN&CD); Group C (routine nutrition advice and oral chlorhexidine decontamination, RN&CD)

SUMMARY:
The goal of this multicenter randomized controlled trial is to explore the efficacy of perioperative oral decontamination and immunonutrition supplement to prevent postoperative pulmonary complications in elderly patients(≥65 years) receiving elective non-cardiac operations. Participants will be either given immunonutrition supplement versus routine nutrition advice, and oral chlorhexidine decontamination versus routine oral care randomly. The two interventions will be compared with control groups separately regarding postoperative pulmonary complications and other outcomes.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, two-by-two factorial randomized controlled trial evaluating the efficacy of immunonutrition supplementation and oral chlorhexidine decontamination. Patients aged 65 years and older who are scheduled for elective non-cardiac surgeries will be recruited. Participants will be excluded if they have contraindication to the intervention. The patients will be randomized into four groups in 1:1:1:1 ratio (oral decontamination vs routine oral care, immunonutrition supplementation vs routine nutrition advice). The primary outcome is the incidence of postoperative pulmonary complications within 7 days after surgery. Secondary outcomes include incidence of pneumonia, infectious complications, comprehensive complication index, postoperative functional recovery, length of hospital stay and hospital expense.

ELIGIBILITY:
Inclusion Criteria:

1. age≥65 years;
2. undergoing major non-cardiac surgery;
3. scheduled for general anesthesia and endotracheal intubation;
4. American Society of Anesthesiologists (ASA) physical status classification I-IV;
5. with intermediate to high risk of respiratory complications assessed by Assess Respiratory Risk in Surgical Patients in Catalonia (ARISCAT) score;
6. informed consent obtained.

Exclusion Criteria:

1. emergency surgery;
2. preoperative pneumonia;
3. allergic to chlorhexidine;
4. severe hepatic/renal dysfunction, incapable of oral feeding, with autoimmune diseases, taking immunosuppressant or immunoregulation medications, or with other contraindication to immunonutrition supplementation;
5. expected intervention of immunonutrition<3 days.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 592 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pulmonary complications | within 7 days after surgery
  composite outcome of postoperative pulmonary complications, including pneumonia, atelectasis, pneumothorax, bronchospasm, pleural effusion, hypoxemia, acute respiratory failure, prolonged mechanical ventilation, unplanned re-intubation,etc.

SECONDARY OUTCOMES:
postoperative pneumonia | within 7days and 30 days after surgery
  defined according to the US Centers for Disease Control Definition
postoperative pulmonary complications | within 30 days after surgery
  composite outcome of postoperative pulmonary complications, including pneumonia, atelectasis, pneumothorax, bronchospasm, pleural effusion, hypoxemia, acute respiratory failure, prolonged mechanical ventilation, unplanned re-intubation,etc.
postoperative infectious complications | within 7days and 30 days after surgery
  composite outcome including surgical site infection, respiratory infection, urinary tract infection, intra-abdominal infection, blood stream infection, etc.
postoperative complications | within 7days and 30 days after surgery
  defined using comprehensive complication index
postoperative recovery | within 7days and 30 days after surgery
  assessed by 15-item quality of recovery questionnaire and WHO disability assessment schedule 2.0
hospitalization expenses | upon hospital discharge, typically 1-2 weeks
  total expense during the hospital stay
length of hospital stay | upon hospital discharge，typically 1-2 weeks
  days of in hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, Dr, Principal Investigator — Peking Union Medical College Hospital
Locations (2):
- China (2):
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Peking Union Medical College Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
All data will be available from the corresponding author upon reasonable request.
Time Frame: 6 months after publication of study results.
Access Criteria: Data will be available from the corresponding author upon reasonable request.

REFERENCES:
- [Derived] Yu J, Che L, Zhu Q, Xu L, Fu J, Zhang Y, You M, Zheng X, Liu C, Huang L, Wang W, Yao L, Fan G, Chen J, Zhang J, Huang Y. Perioperative Oral decontamination and ImmunoNuTrition (POINT) to prevent postoperative pulmonary complications in elderly patients scheduled for elective non-cardiac surgeries: protocol for a multicentre, randomised controlled trial. BMJ Open. 2025 May 14;15(5):e092068. doi: 10.1136/bmjopen-2024-092068. PMID 40374210